CLINICAL TRIAL: NCT00166361
Title: Long-Term Temporary Drainage of Malignant Extrinsic Ureteral Obstruction Secondary to Inoperable Pelvic or Abdominal Malignancies Using the Memokath 051 Ureteral Stent
Brief Title: Drainage of Malignant Extrinsic Ureteral Obstruction Using the Memokath Ureteral Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Pnn Medical A/S (Industry)
Responsible Party: Principal Investigator, Lance A. Mynderse, MD, Consultant in Urology (Surgical), Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 255-03
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-06

CONDITIONS: Ureteral Obstruction
Keywords: Extrinsic ureteral obstruction; Memokath 051 Ureteral Stent; JJ Stent; Stent
MeSH Terms: conditions — Ureteral Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memokath 051 Ureteral Stent (Experimental): Subjects assigned to this arm received a Memokath 051 Ureteral Stent.
  Interventions: Device: Memokath 051 Ureteral Stent
- JJ Stent (Active Comparator): Subjects assigned to this arm received a JJ stent.
  Interventions: Device: JJ Stent

INTERVENTIONS:
Device: Memokath 051 Ureteral Stent — The Memokath 051 ureter stent is used for the treatment of malignant or benign ureteric strictures in both men and women. The stent design consists of a tightly-coiled nickel-titanium alloy, with a diameter of 10.5 French (Fr) and a fluted proximal diameter expanding to 22 Fr. The stent is manufactured in multiple lengths which are chosen to position the device across the narrowed area rather than crossing the ureteropelvic or ureterovesical junction. It has a thermal memory system for its predetermined shape; the stent softens at temperatures below 10 degrees Celsius but regains its shape when heated above 55 degrees Celsius.
  Arms: Memokath 051 Ureteral Stent
Device: JJ Stent — A JJ stent is a flexible plastic tube that drains urine from the kidney to the bladder and is supposed to stay in place temporarily. There is a coil on each end to keep the stent in place, preventing the stent from migrating down and out from the kidney or up from the bladder into the ureter. The stent can stay in place for few weeks to 3 months or more depending on the indication. If left for more than 6-9 months some stents may get encrusted leading to stone formation around the stent.
  Other Names: Double J stent
  Arms: JJ Stent

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Memokath 051 ureteral stent as a long-term temporary and minimally invasive means of providing ureteral drainage in the setting of malignant extrinsic ureteral obstruction secondary to inoperable abdominal or pelvic malignancies. Up to 15 adults who have extrinsic ureteral obstruction secondary to an inoperable abdominal or pelvic malignancy and need ureteral stent drainage will undergo outpatient placement of the ureteral stent. Ongoing monitoring will continue for as long as the stent is in place.

DETAILED DESCRIPTION:
The Memokath 051 ureteral stent is a device designed to provide long-term temporary ureteral drainage in the setting of extrinsic ureteral obstruction secondary to inoperable pelvic and abdominal malignancies or secondary to changes caused by surgery, chemotherapy, or radiation for pelvic and/or abdominal malignancies. The management of malignant extrinsic ureteral obstruction secondary to inoperable neoplastic disease of the abdomen or pelvis is a common urologic problem, and has important implications for a patient's quality as well as quantity of life, which has been estimated to generally range between 6.5 to 23 months in this population. Currently, extrinsic ureteral obstructions are usually managed with double-J ureteral stents, placed either cystoscopically, or antegrade via a percutaneous nephrostomy tube. Double-J stents are prone to encrustation and obstruction over time, necessitating stent exchange under general anesthesia every 3 to 4 months. These repeat surgical procedures under general anesthesia carry subsequent risks of infection, drug reactions, and iatrogenic injury, leading to degradation in the quality of life of these patients who often have a year or less to live. To circumvent these disadvantages, the nickel-titanium Memokath 051 ureteral stent was developed to provide a means of minimally invasive long-term temporary ureteral drainage.

This is a prospective non-randomized clinical study to evaluate the efficacy of the Memokath 051 ureteral stent in managing extrinsic malignant ureteral obstruction secondary to an inoperable abdominal or pelvic malignancy or secondary to changes caused by surgery, chemotherapy, or radiation for pelvic and/or abdominal malignancies. Enrollment of study subjects will take place over a period of two to three years for to a total of 15 patients.

A control group 10 patients with extrinsic ureteral obstruction secondary to an inoperable pelvic or abdominal malignancy or secondary to changes caused by surgery, chemotherapy, or radiation for pelvic and/or abdominal malignancies and treated by other urologic staff surgeons in a standard fashion with retrogradely placed double-J stents will also be followed every 3 to 4 months.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of extrinsic ureteral obstruction

   1. secondary to inoperable pelvic or abdominal malignancy or
   2. secondary to changes caused by surgery, chemotherapy, or radiation for pelvic and/or abdominal malignancies who have had >2 standard double J stent exchanges with no prospect of being stent-free
2. Life expectancy greater than 4 months
3. Adult patient (18 years of age or older)
4. Preoperative medical examination clearing the patient for general anesthesia
5. No active urinary tract infection by urinalysis and urine culture.

Exclusion Criteria:

1. Ureteral obstruction of a benign or intrinsic etiology
2. Lower urinary tract abnormality precluding cystoscopic stent placement
3. Patients with a solitary kidney
4. Patients not willing or unable to receive their post-operative follow-up at the Mayo Clinic in Rochester, Minnesota
5. Pregnant female patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance A Mynderse, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Oncologic practice of the Mayo Clinic, Rochester, Minnesota from February 2004 to May 2011.
Pre-assignment Details: 29 subjects were enrolled, 4 subjects were screen failures, and were not treated, one subject was treated as a compassionate use patient with a smaller memokath stent.
Period: Overall Study
Arm/Group | Memokath 051 Ureteral Stent | JJ Stent
Started | 14 | 10
Completed | 14 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memokath 051 Ureteral Stent | JJ Stent | Total
Number analyzed (Participants) | 14 | 10 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 0 | 9
  >=65 years | 5 | 10 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Stent Dwell Time
Description: Stent dwell time is defined as the amount of time a stent can remain in the body after it placed, before it needs to be removed due to failure.
Time Frame: baseline to 59 months after placement of stent
Measure: Mean (Full Range); unit: months
Arm/Group | Memokath 051 Ureteral Stent | JJ Stent
Number analyzed (Participants) | 14 | 10
months | 17 [1 to 59] | 3.97 [2.56 to 5.36]

ADVERSE EVENTS:
Arm/Group | Memokath 051 Ureteral Stent | JJ Stent
Serious Adverse Events (participants affected / at risk) | 12/14 | 2/10
Other Adverse Events (participants affected / at risk) | 10/14 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memokath 051 Ureteral Stent (N=14) | JJ Stent (N=10)
Surgery related to underlying disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Carcinoid heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure related to underlying disease (Cardiac disorders) | 1 (1) | 0 (0)
Ureteral Obstruction (Renal and urinary disorders) | 7 (7) | 0 (0)
Bowel Obstruction (Gastrointestinal disorders) | 4 (4) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (2) | 0 (0)
Hospitalization due to disease progression (Renal and urinary disorders) | 3 (3) | 0 (0)
Edema of ureter (Renal and urinary disorders) | 2 (2) | 0 (0)
Stent migrated into bladder (Surgical and medical procedures) | 1 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0) — due to bowel obstruction
Acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) — due to bowel obstruction
Stent encrustation/obstruction (Injury, poisoning and procedural complications) | 4 (6) | 0 (0)
Acute Chronic Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hydroureteronephrosis (Renal and urinary disorders) | 3 (3) | 0 (0)
Hospitalization for fractured ankle (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Trouble with stent placement due to faulty guide wire (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Atropy of the kidney (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrectomy (Renal and urinary disorders) | 0 (0) | 1 (1)
Partial ureterectomy (Renal and urinary disorders) | 0 (0) | 1 (1)
Hospitalization for sepsis (General disorders) | 0 (0) | 2 (2)
Hospitalization for urinary tract infection (UTI) (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memokath 051 Ureteral Stent (N=14) | JJ Stent (N=10)
Essential hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Flank pain (Renal and urinary disorders) | 6 (8) | 3 (4)
Groin pain (General disorders) | 3 (3) | 3 (5)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Iliac pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Left lower quadrant pain (General disorders) | 3 (4) | 0 (0)
Right lower quadrant pain (General disorders) | 0 (0) | 1 (3)
Thigh pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acid reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Difficulty eating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (10) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (7) | 0 (0)
Bladder spasms (Renal and urinary disorders) | 0 (0) | 1 (2)
Decreased renal function (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 7 (8) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterectasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary tract infections (UTI) (Renal and urinary disorders) | 9 (19) | 4 (7)
Urine leakage (Renal and urinary disorders) | 0 (0) | 3 (6)
Burning when urinating (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1)
Deydration (General disorders) | 1 (1) | 0 (0)
Fall resulting in fractured ribs (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 3 (4) | 1 (1)
Fever (General disorders) | 3 (4) | 2 (2)
Fragility (General disorders) | 2 (2) | 0 (0)
Headache (General disorders) | 1 (5) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0)
Knee weakness (General disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Night Sweats (General disorders) | 1 (1) | 0 (0)
Weight Loss (General disorders) | 1 (1) | 0 (0)
Tiredness/fatigue (General disorders) | 2 (3) | 0 (0)
Weakness (General disorders) | 2 (2) | 0 (0)
Vasovagal episode (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Low number of subjects in each cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No